CLINICAL TRIAL: NCT06779279
Title: Adjunctive Oral Hygiene Aids in Reducing Commonly Seen Oral Hygiene Parameters Among Orthodontic Patients: a Randomized Controlled Trial
Brief Title: Adjunctive Oral Hygiene Aids in Reducing Oral Hygiene Parameters Among Orthodontic Patients
Acronym: D-F-H-17-Dec
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: sudhir rama varma (Other)
Responsible Party: Sponsor-Investigator, sudhir rama varma, Clinical Assistant Professor, Ajman University
Organization: Ajman University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D-F-H-17-Dec
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Gingival Bleeding; Dental Plaque Accumulation
Keywords: waterflosser; superfloss; gingival bleeding; Dental Plaque
MeSH Terms: conditions — Gingival Hemorrhage; Dental Plaque

STUDY DESIGN:
Intervention Model Description: The study comprised 18-35-year-old girls and boys planning orthodontic treatment. Participants had upper right tooth to lower left molar braces, a pocket depth of 3 mm, and had not flossed in 24 hours. Smoking, periodontal disease, missing teeth, voids between teeth in the arch, and systemic disorders disqualified participants.
Masking Description: No masking done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- water flosser and super flosser (Active Comparator): One side of the mouth was flossed with Super Floss® (Oral-B) and the other with Waterflosser®.
  Interventions: Device: Water flosser and super flosser
- Orthodontic brushes (Active Comparator): One side of the mouth will be brushed with Orthodontic brushes
  Interventions: Device: Orthodontic brush

INTERVENTIONS:
Device: Water flosser and super flosser — Participant will use in one area superfloss and the other area waterfloss
  Arms: water flosser and super flosser
Device: Orthodontic brush — Participant will use orthodontic brush to brush in the upper/lower quadrant
  Arms: Orthodontic brushes

SUMMARY:
Adult orthodontic patients aged 18-30 were included in a randomised, singleblind clinical research using a split-mouth design at a dental clinic. Both theWaterflosser® and the Super-Floss® water flossers are manufactured by Oral-B.

DETAILED DESCRIPTION:
In order to reduce gingival inflammation and remove subgingival plaque, oral hygiene therapy is necessary. The available evidence indicates that mechanical plaque control, which patients administer themselves daily, is the most important factor in managing and reducing plaque accumulation. Aim: This research aimed to determine whether Waterflosser or Superfloss was more effective in lowering the gingival bleeding score and plaque. Methods: Adult orthodontic patients aged 18-30 were included in a randomised, single-blind clinical research using a split-mouth design at a dental clinic. Both the Waterflosser® and the Super-Floss® water flossers are manufactured by Oral- B.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-35 years undergoing orthodontic treatment and
* systemically healthy without habits

Exclusion Criteria:

* Participants not undergoing orthodontic treatment and participants undergoing orthodontic treatment in the included age category but with systemic conditions prevalent
* missing teeth and
* treated previously for periodontal conditions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Gingival Bleeding | Through study completion, an average of 1 month
  Gingival bleeding scores will be evaluted 0-no gingival bleeding
  1. mild gingival bleeding
  2. moderate gingival bleeding
  3. spontaneous gingival bleeding

SECONDARY OUTCOMES:
Number of Participants with Dental Plaque | Through study completion, an average of 1 month
  Dental Plaque scores will be evaluated 0-No dental plaque
  1. Upto 1/3rd of the tooth surface
  2. more than 1/3rd and less than 2/3rd of tooth surface
  3. more than 2/3rd of tooth surface

CONTACTS AND LOCATIONS:
Overall Officials: sudhir Rama Varma, MDS, Principal Investigator — Ajman University
Locations (1):
- Ajman university, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
study protocol, Data and statistical analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Will be available from start of the study till 12 months
Access Criteria: The data will be shared upon request